CLINICAL TRIAL: NCT05613283
Title: Primary Cervical Cancer Screening by Self-sampling HPV Test
Acronym: PREVENT
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: BeijingNewBiorayTechnologyCo.,Ltd. (Unknown); Hangzhou Newhorizon Health Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Wang Jianliu, Chief physician, Peking University People's Hospital
Other Study IDs: NH-3004
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Human Papillomavirus Infection; Cervical Cancer; Negative For Intraepithelial Lesion Or Malignancy; Atypical Squamous Cells of Undetermined Significance; Atypical Squamous Cells, Cannot Rule Out High-grade Squamous Intraepithelial Lesion; Cervical Squamous Intraepithelial Lesion; Low-Grade Squamous Intraepithelial Lesions; High-Grade Squamous Intraepithelial Lesions; Cervical Intraepithelial Neoplasia Grade I; Cervical Intraepithelial Neoplasia Grade II; Cervical Intraepithelial Neoplasia, Grade III; Atypical Glandular Cells; Atypical Glandular Cells Not Otherwise Specified; Atypical Glandular Cells, Favor Neoplastic; Cervical Squamous Cell Carcinoma; Adenocarcinoma in Situ; Cervical Adenocarcinoma
Keywords: Self-sampling HPV testing; Human papilloma virus; Cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Atypical Squamous Cells of the Cervix; Squamous Intraepithelial Lesions; Uterine Cervical Dysplasia; Adenocarcinoma in Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Accuracy verification group: Assessment reagent urine sample HPV-PCR test result Assessment reagent vaginal secretion sample HPV-PCR test result Comparative Methods NGS Nucleic Acid Sequencing Results
- Consistency verification group: Assessment reagent urine sample HPV-PCR test result Assessment reagent vaginal secretion sample HPV-PCR test result ApprovedListed Reagent Cervical Sample HPV-PCR Test Result
- Efficacy and safety verification group: Thin-layer liquid-based cytology (TCT) results panel Colposcopy results Tissue biopsy pathological diagnosis result

SUMMARY:
Cervical cancer seriously threatens women's health and HPV infection is the main cause of cervical cancer. Traditionally, Cervical cancer screening is based on cervical exfoliated cell samples collected by health care provider, which is labor consuming and the coverage and compliance are both relatively low in some areas. Non-invasive hrHPV self-sampling test appears to be more acceptable and may improve the HPV screening coverage. This study aims to evaluate the clinical performance of a newly developed urine/vaginal self-sampling hrHPV test in Cervical cancer screening.

DETAILED DESCRIPTION:
This study is a prospective multi-center clinical trial in China. Eligible participants are cervical cancer screening population who meet the enrollment criterias. All the participants are required to provide urine and vaginal samples by self-sampling, as well as the cervical exfoliated cell samples (by HCP). Participants may undergo colposcopy examination depending on the test results, and they will be followed up for three years.

The high-risk human papillomavirus nucleic acid detection kit (PCR-fluorescent probe method) developed by New Horizon Co., Ltd . is suitable for in vitro qualitative detection of 14 types of high-risk HPV ( 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68) nucleic acid.

The clinical performance of the self-sampling test will be assessed base on the following outcomes:

1. The sensitivity for detecting CIN2+
2. The specificity in non-CIN2+ population
3. The risk of developing CIN2+ in test positive cohort and test negative cohort
4. The accuracy of detecting hrHPV

ELIGIBILITY:
Inclusion Criteria:

* a. Females aged 21-65; b. have a history of sexual life; c. The patients were voluntarily enrolled and signed the informed consent.

Exclusion Criteria:

* Accuracy Verification:

Subjects meeting any of the following criteria will be excluded:

1. Known pregnant subjects.
2. Participants who have undergone total hysterectomy.
3. Participants who have received cervical resection therapy or ablative therapy within 12 months, such as cryo, laser, microwave, coagulation, cryotherapy, LEEP, large loop electrosurgery (LLETZ), cold knife conization (CKC), laser conization, or ablation.
4. Participants with poor compliance or researchers who believe that they are not suitable to participate in this study.

   * Primary screening use:

Subjects meeting any of the following criteria will be excluded:

1. Known pregnant subjects.
2. Participants who have undergone total hysterectomy.
3. Participants who have received cervical resection therapy or ablative therapy within 12 months, such as cryo, laser, microwave, coagulation, cryotherapy, LEEP, large loop electrosurgery (LLETZ), cold knife conization (CKC), laser conization, or ablation.
4. Those with known history of cervical cancer.
5. Participants who participated in cervical cancer screening programs or underwent cervical cytology within 12 months.
6. Participants with poor compliance or researchers who believe that they are not suitable to participate in this study.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on biological sex
Study Population: The population of clinical validity verification is all screening population, that is, women who need to undergo routine cervical cancer screening and the results of cervical cytology are unknown; Accuracy verification needs to include part of the screening population and part of the outpatient population, that is, women who intend or need to undergo colposcopy or cervical cancer screening for clinical visits.
Sampling Method: Non-Probability Sample
Enrollment: 17875 (Estimated)
Dates: Start 2022-11-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy verification | 2023/12
  Calculate the positive coincidence rate, negative coincidence rate, total coincidence rate, and Kappa value of the comparison reagents and calculate the 95% confidence interval to verify the accuracy of detecting HPV infection.
Clinical validity verification | 2027/06
  The consistency of HPV detection of different sample types was analyzed, and the absolute risk value, relative risk value and 95% confidence interval of the development of ≥CIN2 in different primary screening types were calculated and used to verify the safety and effectiveness of the intended use of cervical cancer primary screening.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Background] Nelson EJ, Maynard BR, Loux T, Fatla J, Gordon R, Arnold LD. The acceptability of self-sampled screening for HPV DNA: a systematic review and meta-analysis. Sex Transm Infect. 2017 Feb;93(1):56-61. doi: 10.1136/sextrans-2016-052609. Epub 2016 Oct 19. PMID 28100761
- [Background] Bruni L, Albero G, Serrano B, et al.ICO/IARC Information Centre on HPV and Cancer (HPV Information Centre). Human Papillomavirus and Related Diseases in China. Summary Report 22 October 2021. [EB/OL].www.hpvcentre.net
- [Background] Wu RF, Du H. [Development of model based on self-sampling HPV testing for cervical cancer screening]. Zhonghua Fu Chan Ke Za Zhi. 2017 Sep 25;52(9):582-585. doi: 10.3760/cma.j.issn.0529-567X.2017.09.002. No abstract available. Chinese. PMID 28954445
- [Background] Bernal S, Palomares JC, Artura A, Parra M, Cabezas JL, Robles A, Martin Mazuelos E. Comparison of urine and cervical samples for detecting human papillomavirus (HPV) with the Cobas 4800 HPV test. J Clin Virol. 2014 Dec;61(4):548-52. doi: 10.1016/j.jcv.2014.10.001. Epub 2014 Oct 12. PMID 25453566
- [Background] Hagihara M, Yamagishi Y, Izumi K, Miyazaki N, Suzuki T, Kato H, Nishiyama N, Koizumi Y, Suematsu H, Mikamo H. Comparison of initial stream urine samples and cervical samples for detection of human papillomavirus. J Infect Chemother. 2016 Aug;22(8):559-62. doi: 10.1016/j.jiac.2016.05.009. Epub 2016 Jun 21. PMID 27342077
- [Background] Pathak N, Dodds J, Zamora J, Khan K. Accuracy of urinary human papillomavirus testing for presence of cervical HPV: systematic review and meta-analysis. BMJ. 2014 Sep 16;349:g5264. doi: 10.1136/bmj.g5264. PMID 25232064
- [Background] Combita AL, Gheit T, Gonzalez P, Puerto D, Murillo RH, Montoya L, Vorsters A, Van Keer S, Van Damme P, Tommasino M, Hernandez-Suarez G, Sanchez L, Herrero R, Wiesner C. Comparison between Urine and Cervical Samples for HPV DNA Detection and Typing in Young Women in Colombia. Cancer Prev Res (Phila). 2016 Sep;9(9):766-71. doi: 10.1158/1940-6207.CAPR-16-0038. Epub 2016 Jul 14. PMID 27417431
- [Background] Cho HW, Shim SR, Lee JK, Hong JH. Accuracy of human papillomavirus tests on self-collected urine versus clinician-collected samples for the detection of cervical precancer: a systematic review and meta-analysis. J Gynecol Oncol. 2022 Jan;33(1):e4. doi: 10.3802/jgo.2022.33.e4. Epub 2021 Oct 7. PMID 34783207
- [Background] Arbyn M, Verdoodt F, Snijders PJ, Verhoef VM, Suonio E, Dillner L, Minozzi S, Bellisario C, Banzi R, Zhao FH, Hillemanns P, Anttila A. Accuracy of human papillomavirus testing on self-collected versus clinician-collected samples: a meta-analysis. Lancet Oncol. 2014 Feb;15(2):172-83. doi: 10.1016/S1470-2045(13)70570-9. Epub 2014 Jan 14. PMID 24433684
- [Background] Camara H, Zhang Y, Lafferty L, Vallely AJ, Guy R, Kelly-Hanku A. Self-collection for HPV-based cervical screening: a qualitative evidence meta-synthesis. BMC Public Health. 2021 Aug 4;21(1):1503. doi: 10.1186/s12889-021-11554-6. PMID 34348689
- [Background] Belinson JL, Wang G, Qu X, Du H, Shen J, Xu J, Zhong L, Yi J, Yi X, Wu R. The development and evaluation of a community based model for cervical cancer screening based on self-sampling. Gynecol Oncol. 2014 Mar;132(3):636-42. doi: 10.1016/j.ygyno.2014.01.006. Epub 2014 Jan 14. PMID 24440471
- [Background] Xu H, Yu Y, George W, Smith JS, Hu S, Dang L, Zhang X, Pan Q, Qiao Y, Zhao F. Comparison of the performance of paired urine and cervical samples for cervical cancer screening in screening population. J Med Virol. 2020 Feb;92(2):234-240. doi: 10.1002/jmv.25597. Epub 2019 Sep 30. PMID 31535725
- [Background] Belinson JL, Hu S, Niyazi M, Pretorius RG, Wang H, Wen C, Smith JS, Li J, Taddeo FJ, Burchette RJ, Qiao YL. Prevalence of type-specific human papillomavirus in endocervical, upper and lower vaginal, perineal and vaginal self-collected specimens: Implications for vaginal self-collection. Int J Cancer. 2010 Sep 1;127(5):1151-7. doi: 10.1002/ijc.25144. PMID 20039323
- [Background] 毛康娜, 刘艳欣, 陶惠芬.14398名妇女宫颈癌筛查结果分析[J]. 河南医学研究,2021,30(16):2921-2923.